CLINICAL TRIAL: NCT04760041
Title: Nebulized Midazolam vs. Oral Midazolam as a Sedative Premedication in Pediatric Anesthesia: A Randomized Comparative Study
Brief Title: Nebulized vs. Oral Midazolam Sedation in Pediatric Anesthesia: A Randomized Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Mohamed Abd El Moneim Soaida, MD, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SMS2021-1
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Preoperative Sedation
MeSH Terms: interventions — Nebulizers and Vaporizers; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nebulized midazolam group (Active Comparator): 36 children will receive nebulized midazolam 0.2 mg/kg in 3 ml normal saline plus 5 ml clear juice 30 min before undergoing general anesthesia
  Interventions: Drug: Midazolam nebulized
- oral midazolam group (Active Comparator): 36 children will receive oral midazolam 0.5 mg/kg in 5 ml clear juice plus nebulizer of 3 ml normal saline 30 min before undergoing anesthesia
  Interventions: Drug: Midazolam oral solution

INTERVENTIONS:
Drug: Midazolam nebulized — midazolam nebulized
  Other Names: nebulizer
  Arms: nebulized midazolam group
Drug: Midazolam oral solution — midazolam given oral
  Other Names: oral
  Arms: oral midazolam group

SUMMARY:
This study is to be carried out to compare nebulized and oral midazolam in achievement of a satisfactory level of sedation, Ramsey Sedation Score (RSS) of 4, within 30 mins of midazolam administration in pediatrics.

DETAILED DESCRIPTION:
This study is to be carried out to compare nebulized midazolam and oral midazolam in achievement of a satisfactory level of sedation, Ramsey Sedation Score (RSS) of 4, within 30 mins of midazolam administration in pediatric surgical patients.

In Pediatric Specialized Hospital, Cairo University 72 pediatric patients scheduled for undergoing general or uro-surgical operations under general anesthesia will be included in this double-blinded study. Patients will be randomly assigned into two equal groups, each group including 36 patients. In one group 36 children will receive nebulized midazolam 0.2 mg/kg in 3 ml normal saline plus 5 ml clear juice (orally) 30 min before undergoing general anesthesia. In the other group 36 children will receive oral midazolam 0.5 mg/kg in 5 ml clear juice plus nebulizer of 3 ml normal saline 30 min before undergoing GA.

level of sedation will be compared between both groups

ELIGIBILITY:
Inclusion Criteria:

* Patients from 2 to 6 years undergoing uro-surgery and general surgical procedures.
* Duration of surgery 1-2 hours
* Gender eligible for the study: both.
* ASA I-II.

Exclusion Criteria:

* ASA III-IV
* Patients with elevated levels of serum ALT, Creatinine.
* Emergency surgeries.
* Pre-existing neurologic disease.
* Parent refusal.
* History of allergy to midazolam.
* Patients with atopy or a history of asthma.
* Lengthy procedures of more than 2 hours

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Time required to reach a satisfactory level of sedation | from time of applying the nebulizer until 30 minutes
  time to reach ramsay sedation score 4

SECONDARY OUTCOMES:
Acceptability of method of administration of midazolam by a grading system | from time of giving midazolam oral or nebulized till 30 minutes
  Facemask acceptance will be graded as poor (terrified, crying, and combative),fair (moderate fear of mask not calmed with reassurance),good (slight fear of mask, easily reassured), or excellent (unafraid, cooperative, and accepts mask readily).
Ease of separation from parents | from 30 minutes after receiving midazolam till transfer to operating room
  using ease of separation and induction scoring system:
  1. Excellent: patient unafraid, cooperative, or asleep
  2. Good: slight fear and/or crying, quiet with reassurance
  3. Fair: moderate fear and crying, not quiet with reassurance
  4. Poor: crying, need for restraint
acceptability of Face mask by grading systen | from time of applying face mask till time of getting asleep at 1 minute intervals
  Facemask acceptance was graded as poor (terrified, crying, and combative), fair (moderate fear of mask not calmed with reassurance), good (slight fear of mask, easily reassured), or excellent (unafraid, cooperative, and accepts mask readily)
Recovery time | time from discontinuation of anesthesia until regaining baseline sedation score at 5 minute intervals
  time to recover
Changes in mean arterial blood pressure | from start of sedation till 1 hour postoperative at 5 minute intervals
  Changes in mean arterial blood pressure measured in mmHg
changes in oxygen saturation | from start of sedation till 1 hour postoperative at 5 minute intervals
  changes in oxygen saturation
changes in heart rate | from start of sedation till 1 hour postoperative at 5 minute intervals
  changes in heart rate
  changes in heart rate (beats per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided